CLINICAL TRIAL: NCT05860517
Title: Translation and Cultural Adaptation of Caregiver Priorities and Child Health Index of Life With Disability (CPCHILD)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RIPHAH/RCRS/REC/Letter-01269
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Caregiver Priorities and Child Health Index; CPCHILD; Cultural validation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a tool translation an validation study. CPCHILD will be translated in Urdu language and it's translated version will be validated. Translated version's reliability and validity will also be assessed. The WHO guidelines for tool translation study will be followed.

DETAILED DESCRIPTION:
Phase 1: Translation Translation of English version of CPCHILD into Urdu version will be done according to the WHO guidelines.

Step I: Forward translation (one way) into target language:

A linguistic expert with bilingual (English and Urdu) expertise will translate the original English version into Urdu.

Step II: Synthesis:

An independent bilingual translator will then compare the translated version (Urdu) with the original version (English) of the instrument.

Step III: Blind Backward translation:

A blinded backward translation of initially translated version will be done. Bilingual expert with preferably having Urdu as his/her mother language will be blinded to original version, will translate Urdu version into English.

Step IV: Pretesting:

10 subjects including translators, physical therapists and researchers will fill out the questionnaire before submission of final version.

Step V: Expert (multidisciplinary) committee review:

An expert committee including translators, researchers, and health care practitioner would develop a pre-final version after reviewing all the translations.

Phase 2: Psychometric testing Full psychometric testing of the CPCHILD in individuals from the target population to revise and refine the items according to instructions and guidelines of the final version of the questionnaire in the target language as well as to establish internal consistency reliability, test-retest reliability, homogeneity, construct-related validity, criterion-related validity, factor structure, and model fit of the instrument. Data will be collected from patients on both scales to assess for validity, reliability and psychometric properties.

Reliability In the present study, the reliability of the CPCHILD will be determined by assessing test-retest reliability across repeated measures and internal consistency.

Test-retest reliability:

For test-retest reliability, the scale will be completed once a day by the same participant who keeping the same signs and symptoms. A time interval of 1 week will be allowed between the assessments. Intra class correlation coefficient (ICC) will be used to evaluate test- retest reliability.

Internal consistency:

Internal consistency is a measure of the extent to which items in a both scales are correlated (homogeneous), thus measuring the same concept.

Cronbach's alpha will be calculated to determine the internal consistency.

Content validity:

Content validity is the degree to which the content of an instrument has an adequate reflection of the construct being measured. Content validity will be assessed by determining the completeness of item responses.

Construct validity:

Construct validity refers to the extent to which scores on a particular instrument relate to other measures in a way that is consistent with theoretically derived hypotheses concerning the concepts that are being measured. Construct validity will be investigated using concurrent validity. Construct validity will be assessed by measuring the correlation between CPCHILD scale and child health questionnaire. Spearman and Pearson correlation coefficients would be calculated for determining validity.

Phase 3:

A survey would be done to assess the level of disability and health status of cerebral palsy through CPCHILD questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with cerebral palsy
* Age 3 to 15 years
* Gross motor function score II, III, IV

Exclusion Criteria:

* Cognitive, visual or hearing impairment
* Any comorbidity or metabolic disorders

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosed cases of Cerebral palsy who fulfill the inclusion criteria with gross motor function level II, III, IV.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Caregiver priorities and child health index of life with disability (CPCHILD) | Baseline (one time assessment)
  Priorities of caregivers along with level of health status of the Cerebral Palsy child. The score ranges from 0 to 100, 0 is the best and 100 is worst.
Health Related Quality of Life (HRQoL) | Baseline (one time assessment)
  The tool is used to determine the quality of life and health status of subjects. The score ranges from 0 to 100, lower scores indicate better outcome and higher scores indicate worse outcome.
International physical activity questionnaire (IPAQ) | Baseline (one time assessment)
  International physical activity questionnaire (IPAQ) is used to determine the level of physical activity in certain population. The subjects may have the levels as; inactive, minimal active, moderate and highly active depending on the scores.
Health related quality of life (HRQoL) | Baseline (one time assessment)
  Health related quality of life (HRQoL) will be used to determine the quality of life in subjects with cerebral palsy
Pittsburgh Sleep questionnaire | Baseline (one time assessment)
  Pittsburgh Sleep questionnaire will be use to detrmine the quality of sleep in cerebral palsy subjects.
Trunk impairment scale | Baseline (one time assessment)
  Trunk impairment scale is used for trunk control. The lower the trunk control, the higher chances of disability in cerebral palsy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khushnood, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No